CLINICAL TRIAL: NCT05003895
Title: Phase I Study of GPC3 Targeted CAR-T Cell Therapy in Advanced GPC3 Expressing Solid Tumor Malignancies
Brief Title: GPC3 Targeted CAR-T Cell Therapy in Advanced GPC3 Expressing Hepatocellular Carcinoma (HCC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210030; 21-C-0030
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05-20

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Metastatic Hepatocellular Carcinoma
Keywords: immuno therapy; Targeted Therapy; Leukapheresis; Gene Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Cyclophosphamide; Immunotherapy, Adoptive; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Arm 1 (Experimental): Escalating doses of CAR-T cells
  Interventions: Drug: Cyclophosphamide; Biological: CAR-T cell; Drug: Fludarabine
- 2/ Arm 2 (Experimental): MTD of CAR-T cells
  Interventions: Drug: Cyclophosphamide; Biological: CAR-T cell; Drug: Fludarabine

INTERVENTIONS:
Drug: Cyclophosphamide — Daily x 3 doses on Day -3, -2, -1 300 mg/m2 IV infusion (200 mg/m^2 in Dose Level -1)
Biological: CAR-T cell — Single infusion on Day 0
Drug: Fludarabine — Daily x 2 doses on Day -2 and -1 30 mg/m^2 IV infusion administered following cyclophosphamide

SUMMARY:
Background:

A new cancer treatment takes a person s own T cells, modifies them in a laboratory so they can better fight cancer cells, and then gives them back to the person. Researchers want to see if this treatment can help people with a certain type of liver cancer.

Objective:

To see if a personalized immune treatment, anti-GPC3 CAR-T cells, is safe.

Eligibility:

Adults aged 18 years and older who have Glypican-3 (GPC3) positive HCC, a type of liver cancer.

Design:

Participants will be screened with the following:

Blood and urine tests

Medical history

Physical exam

Heart function tests

Review of their symptoms and their ability to perform their normal activities

Tumor biopsy

Imaging scan of the chest, abdomen, and pelvis

Participants will have leukapheresis. They may have an IV (intravenous catheter, a small tube put into an arm vein) inserted into each arm or get a central line. Blood will be removed. A machine will separate the white blood cells from their blood. The rest of their blood will be returned to them.

Participants will be admitted to the hospital for about 2 weeks. They will get the chemotherapy drugs fludarabine and cyclophosphamide by IV for 3 days. Then they will receive the modified white blood cells by IV.

Participants will have frequent blood draws. They will give blood and tumor samples for research.

Participants will have follow-up visits for the next 15 years. Then they will be contacted by email or phone for the rest of their life. If their disease does not get worse after 5 years, they will continue to be invited to do imaging studies every 6 months.

DETAILED DESCRIPTION:
Background:

* Hepatocellular carcinoma (HCC) is the fifth most common cancer worldwide and the second leading cause of cancer-associated mortality with an average life expectancy of 6-9 months
* Despite the success of several studies showing efficacy in treating HCC, most clinical trials have failed to prove a survival advantage.
* Adoptive T-cell therapy exploits the natural ability of T-cells to recognize and eliminate their target.
* GPC3 is a cell surface protein that is expressed in nearly all HCC yet is undetectable in normal adult hepatic tissues.
* GPC3 is also expressed strongly in some non-HCC solid tumor malignancies.
* We want to evaluate the role of GPC3 targeted chimeric antigen receptor (CAR)-T cells in advanced GPC3 expressing HCC as well as other advanced solid tumor malignancies with GPC3 expression.

Objective:

-To determine the safety and feasibility of T-cells, expressing a novel humanized anti-GPC3 chimeric antigen receptor, in participants with advanced solid tumor malignancy, expressing GPC3.

Eligibility:

* Histologically confirmed diagnosis of hepatocellular carcinoma or other solid tumor malignancy.
* GPC3 positivity of >= 25% by immunohistochemistry
* At least 1 measurable lesion by RECIST v 1.1 criteria
* Age >= 18 years

Design:

* We plan to conduct a phase I dose escalation designed clinical trial using CAR (hYP7)-T cells in participants with advanced hepatocellular carcinoma or other advanced solid tumor malignancy, expressing GPC3.
* Participants will undergo leukapheresis
* Participants will receive a lymphocyte depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused CAR-expressing T cells
* Following the T cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* The participants will be closely monitored during the first year after cell infusion and followed for life.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histopathological confirmation of HCC or other solid tumor malignancy by the NCI Laboratory of Pathology
* Participants must:

  * have progressed on at least 1 prior line of treatment

OR

--been intolerant of at least 1 prior line of treatment.

* Participants must have at least 1 focus of disease that is amenable to mandatory tumor biopsy prior to study treatment initiation to determine tumor GPC3 expression and be willing to undergo this. Ideally, the biopsied lesion should not be one of the target measurable lesions, although this can be up to the discretion of the investigators.
* Tumor must have GPC3 positivity of >= 25% by immunohistochemistry on freshly collected biopsy
* Participants must have at least 1 measurable lesion by RECIST version 1.1
* Participants must have a disease that is not amenable to potentially curative resection, ablation, or transplantation.
* Age >= 18 years.
* Performance status (ECOG) 0-1
* Participants must have adequate organ and marrow function as defined below:

ANC: >= 1,000/mcL

Platelets: >= 75,000/mcL

Hemoglobin: >= 8 g/dL

total bilirubin: If cirrhosis present: Part of Child Pugh requirement

If no cirrhosis: bilirubin should be <= 1.5 x ULN

ALT or AST: <= 5 x ULN.

Creatinine OR Measured or calculated creatinine clearance (CrCl) (eGFR may also be used in place of CrCl) (A): < 1.5x institution upper limit of normal OR >= 50 mL/min/1.73 m^2 for participant with creatinine levels, >= 1.5 X institutional ULN

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);

AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

(A)Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.

* Normal cardiac ejection fraction (>= 50% by echocardiogram) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 4 weeks before treatment initiation.
* Room air oxygen saturation of 92% or greater.
* Treatment-related toxicities must be resolved to <= grade 1.
* For participants with brain metastases: Participants with <=3 (three or fewer) brain metastases that have been treated with surgery or stereotactic radiosurgery or other form of treatment are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month before protocol treatment.
* The study drugs are harmful to developing human fetus. For this reason, women of childbearing potential must agree to use highly effective contraception (hormonal, intrauterine device (IUD), abstinence, surgical sterilization) at the study entry and up to 12 months after the last dose of combined chemotherapy. Men must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and up to 4 months after the last dose of study drugs. We also recommend men with partners of childbearing potential ask their partners to be on highly effective birth control (hormonal, IUD, surgical sterilization). Men must not freeze or donate sperm within the same period.
* HBV infected participants must be on antivirals and have HBV DNA < 100IU/mL. HCV infected participants can be enrolled with close HCV RNA level monitoring.
* Participants must be able to understand and be willing to sign a written informed consent.
* For participants that do not have a legally authorized representative in place, one must be identified before study treatment starts

Exclusion Criteria

* Prior systemic therapy, an investigational therapy, radiation, and/or surgery within 2 weeks prior to treatment initiation.
* Prior administration of anti-PD-1 or anti-PD-L1 antibodies or other agents that in the opinion of the PI can stimulate immune activity and interfere with an infusion of CAR-T cells within 8 weeks prior to treatment initiation.
* Child-Pugh class B or C liver function
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Note: Participants with a history of abnormal pulmonary function tests but stable obstructive or restrictive pulmonary disease may be eligible per PI discretion.

* Any form of primary immunodeficiency (e.g. severe combined immunodeficiency).
* HIV-positive participants are excluded because HIV causes complicated immune deficiency and study treatment can pose more risks for these participants.
* Participants receiving systemic steroids >= 0.5 mg prednisone equivalent/kg/day. Steroid creams, ointments, and eye drops are allowed. Dose adjustment or discontinuation of medication must occur at least 24 hours prior to conditioning chemotherapy. Use of CART cell therapy in autoimmune diseases has the potential to be associated with serious safety risk. Given that this is an evolving area of research, caution should be exercised and any decision to include participants with autoimmune diseases should be made on a case-bycase basis.
* History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.
* Hospitalization within 7 days prior to treatment initiation.
* Pregnant women are excluded from this study because study therapy can cause fetal harm. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with study therapy, breastfeeding should be discontinued if the mother is treated with study drugs.
* Participants who received live or attenuated vaccine or virus-based vaccine within 30 days before initiation of study therapy
* Participants with a history of seizure disorder
* Participants with an expected life expectancy of less than 3 months before initiation of study therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and feasibility of T-cells, expressing a novel humanized anti-GPC3 chimeric antigen receptor, in participants with advanced solid tumor malignancy, expressing GPC3. | 15 years
  Safety will be reported based on DLTs per dose level as well as reporting specific grades and types of toxicity encountered. Feasibility will be reported descriptively as the fraction of participants overall and per dose level who are able to receive sufficient CAR T cells as required for the specified dose level

SECONDARY OUTCOMES:
To characterize overall survival (OS) | death
  Kaplan-Meier curve and 95% confidence interval for the median OS
To determine the best overall response (BOR) rate according to Response Evaluation Criteria (by RECIST v 1.1) of treatment with T-cells, expressing a novel humanized anti-GPC3 chimeric antigen receptor in participants with advanced HCC, expressi... | every 2-month for the first year, every 3 month for the second year, every 4 month for the third year, and every 6 month afterward until disease progression
  BOR rate will be reported among the 12 participants at the final dose level, along with a 95% two-sided confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0030.html